CLINICAL TRIAL: NCT03047694
Title: Contribution of a Semantic Therapy on a Tactile Tablet in the Alzheimer's Disease, Early and Late Onset
Brief Title: A Lexico-semantic Program on Tactile Tablet for Patients With Alzheimer's Disease
Acronym: SemantiMATT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P140707; 2015-A01312-47 (Other: IDRCB)
Record Dates: First submitted 2016-12-23; First posted 2017-02-09 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Alzheimer Disease
Keywords: Lexico-semantic stimulation; tactile tablet
MeSH Terms: conditions — Alzheimer Disease | interventions — Speech Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tablet group (Experimental): Patients will continue their usual care (1 or more sessions of weekly speech therapy) and will benefit from the therapy on tablet for 3 months.
  Interventions: Other: tablet therapy
- Control group (Active Comparator): Patients will continue their usual care (1 or more sessions of weekly speech therapy)
  Interventions: Other: usual care

INTERVENTIONS:
Other: tablet therapy — stimulation of the lexico semantic system on a tactile tablet therapy for 3 months
  Other Names: Experimental Arm
  Arms: Tablet group
Other: usual care — speech therapy
  Other Names: speech therapy
  Arms: Control group

SUMMARY:
Lexical semantic disorders are described in Alzheimer's disease, and their incidence in everyday life is important to the extent that these disorders affect expression and comprehension.

Providing a tactile tablet stimulation, independent and complementary to speech therapy, could help to maintain certain abilities and reinforce the feeling of autonomy of the patients.

DETAILED DESCRIPTION:
It is a monocentric, controlled, randomized, parallel-group, single-blind clinical trial.

For each of the two forms of Alzheimer's Disease (young or late), it compares two groups of patients: a group benefiting from a tactile tablet semantic stimulation (tablet group) and a control group All patients benefit from a clinical evaluation and a language assessment at M0, M3 and M6. The analyzes will be conducted in intention to treat.

The main criterion is the 3-month variation of the Lexis 3 subtests scores. The two groups will be compared by the Student test.

The number of subjects required is based on the following assumptions: a 10% increase over three months of the Lexis subtests scores in the tablet group and a stability of the scores in the control group. The standard deviation of the variation is assumed to be identical in both groups and equal to 13% at the most. Three scores being compared, tests will be conducted at the 1.67% threshold (Bonferroni correction) to ensure a 5% overall risk of first species. The inclusion of 36 patients in each of the two treatment groups will give 80% power to the study.

ELIGIBILITY:
Inclusion Criteria:

1. Major Patient
2. Patient with a diagnosis of Alzheimer's disease according to DSM-IV and NINCDS-ADRDA criteria.
3. Patient at a moderate stage of the disease: Score at CDR (Clinical Dementia Rating Scale) between 0.5 inclusive and 2 inclusive and MMS score greater than or equal to 10 and lower strictly at 27
4. Lexical-semantic disorder
5. Treatment with pro-cognitive drugs at stable doses for at least 3 months,
6. Speech therapy in progress (2 or 3 sessions per week)
7. Patient with free and informed consent
8. Affiliated to the Health care system
9. Native french speaker,
10. Attendance of a caregiver.

For the early onset group, patients should have started the disease before 65 years of age. The randomization will be stratified according to age (<65 years or> 65 years), enabling to include 2 groups of identical size of young AD (Alzheimer Disease) and Late (Alzheimer Disease) patients, each half distributed in the tablet or control group.

Exclusion Criteria:

1. Other known neurological disease or general illness or major psychic problems that may interfere with cognitive functioning,
2. Patient under guardianship or curatorship
3. Confusion,
4. Cerebral MRI (or scanner for contraindication to MRI), obtained in the context of routine care compatible with a pathological process other than that related to Alzheimer's disease. A discrete or moderate leukoaraiosis (stages 1 and 2 of Fazekas) will not be considered as a criterion of non-inclusion.
5. Uncorrected hearing or visual impairment
6. Inclusion in another intervention protocol.
7. Participation in an additional stimulation workshop

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
variation of performance on naming subtest of the LEXIS | variation from baseline at 3 month
variation of performance on designation subtest of the LEXIS | variation from baseline at 3 month
variation of performance on semantic matching subtest of the LEXIS | variation from baseline at 3 month

SECONDARY OUTCOMES:
variation of performance on DO80 lexico-semantic test | variation from baseline at 3 month and 6 month
variation of performance on verbal fluency lexico-semantic test | variation from baseline at 3 month and 6 month
variation of performance on verbal discrimination of BADAE | variation from baseline at 3 month and 6 month
variation of performance on episodic memory test (RL/RI) | variation from baseline at 3 month and 6 month
variation of performance on Mini-Mental State Examination (MMSE) | variation from baseline at 3 month and 6 month
variation of score on depression scale (HAD) | variation from baseline at 3 month and 6 month
variations on care giver's questionary | variation from baseline at 3 month and 6 month
variation of performance on naming subtest of the LEXIS | variation from 3 month at 6 month
variation of performance on designation subtest of the LEXIS | variation from 3 month at 6 month
variation of performance on semantic matching subtest of the LEXIS | variation from 3 month at 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Agnès MICHON, MD, Principal Investigator — Assistance Publique Hoptiaux de Paris
Locations (2):
- France (2):
  - Hôpital Pitié-Salpêtriere, Paris
  - APHP - Pitié-Salpêtrière Hospital, Paris